CLINICAL TRIAL: NCT05714813
Title: Circuit Resistance Training and Retinal Vascular Changes in Older Persons
Brief Title: Circuit Training and Retina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210271
Record Dates: First submitted 2022-12-21; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Impairment, Progressive; Cerebral Small Vessel Diseases
Keywords: Circuit Resistance Training; High-velocity Training; Retinal Microvasculature; Cognitive Function
MeSH Terms: conditions — Cognitive Dysfunction; Cerebral Small Vessel Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Speed Circuit Resistance Training Group (Experimental): Participants in this group will receive high-speed circuit resistance training 3 times a week for 24 consecutive weeks for a total of 72 training sessions.
  Interventions: Behavioral: High-Speed Circuit Resistance Training
- Control Group (Other): Participants in this arm will receive two lectures on fitness, diet, or cognition each month for 24 weeks for a total of 12 lectures.
  Interventions: Behavioral: Lecture on Diet, Exercise and Cognition

INTERVENTIONS:
Behavioral: High-Speed Circuit Resistance Training — Performance of 24 weeks of high-speed concentric and low-speed eccentric lift across three circuits on eleven pneumatic machines. Each training session will be in person and will last between 45 minutes and one hour.
  Arms: High-Speed Circuit Resistance Training Group
Behavioral: Lecture on Diet, Exercise and Cognition — Lectures on diet, exercise, and cognition. Lectures will be provided in person or online and will last approximately one hour.
  Arms: Control Group

SUMMARY:
The purpose of this research study is to see if high-speed weight training performed in a circuit (using one machine after another) can improve participant heart and brain function, strength, and power in older persons.

ELIGIBILITY:
Inclusion Criteria:

1. 65-90 years of age;
2. Montreal Cognitive Assessment (MoCA) > 23
3. no memory loss complaints

Exclusion Criteria:

1. Uncontrolled cardiovascular or neuromuscular diseases that prevent participation in a training program;
2. Cerebrovascular disease;
3. Malignancy within the previous 5 years;
4. Documented HIV infection or other immunodeficiency syndrome;
5. Any systemic inflammatory or autoimmune conditions such as rheumatoid arthritis, systemic lupus erythematosus, or other serious concomitant medical illness;
6. A history of ocular surgeries (except for cataract surgery more than 6 months ago) or other ocular diseases;
7. Bilateral moderate or severe cataracts;
8. Refractive errors of myopia, hyperopia and/or astigmatism more than 6.0 Diopters.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in retinal vessel density as measured by Optical Coherence Tomography Angiography (OCTA) | Baseline, 24 weeks
  OCTA uses a special camera system and software to measure the densities of the small vessels (microvasculature) of the retinal layers of the eye.

SECONDARY OUTCOMES:
Change in Event Memory as measured by the Picture Sequence Memory Test | Baseline, 24 weeks
  The Picture Sequence Memory Test (PSMT) can test how well a subject can remember events. The participants are asked to recall the sequence of pictures presented over two learning trials. Participants are given credit for each adjacent pair of pictures they correctly put in place. The minimum score is 0 and the maximum score is 17. The higher the score indicates better sequential memory. The test takes approximately seven minutes to administer.
Change in Information Sorting as measured by the NIH List Sorting Test | Baseline, 24 weeks
  The National Institute of Health (NIH) List Sorting Test measures a person's ability to store information for a short time while doing other tasks. It asks the subject to sort and put in order lists of both sounds and pictures. The lists may include animals to be sorted by size, foods to be sorted by size, or a combination of the two to be sorted by size. The minimum score is 0 and the maximum score is 26. A higher score indicates better working memory. The test takes about 7 minutes.
Change in Reaction Time for a Mental Task as measured by the NIH Pattern Comparison Processing Speed Test | Baseline, 24 weeks
  The Pattern Comparison test measures the subject's reaction time and how long it takes the subject to do a mental task. During the test, the subject will be asked to decide whether two visual patterns are the "same" or "not the same." The minimum score is 0 and the maximum score is 130. A higher score indicates better processing speed. The test takes 85 seconds.
Change in Dynamic Balance as measured by the Timed Up-and-Go test | Baseline, 24 weeks
  The Timed Up and Go test (TUG) measures dynamic balance, leg strength and walking speed. For this test the subject will sit back in a chair with the hands in the lap. On go, the subject will get up, walk around a cone that is about 9 feet from the chair, walk back and sit back down. The subject will have one practice trial and two real trials. Healthy individuals between 60 and 80 years of age are expected to complete the TUG in 10 seconds or less. Lower scores indicate a better performance.
Change in the Ability to perform Daily Activities as measured by the Physical Performance Test | Baseline, 24 weeks
  The Physical Performance Test tests daily skills. The subject is asked to write a sentence, pick up some beans from a table and put them in a coffee can, move a book from a table to a shoulder-high shelf, put on and take off a coat, pick up a penny from the floor, turn around 360 degrees, walk 50 feet, and climb up and down some flights of stairs. The minimum score is 0 and the maximum score is 36. A higher score indicates better ability to do daily activities. The test takes about 5 minutes.
Change in Recall and Recognition as measured by the Hopkins Verbal Learning Test | Baseline, 24 weeks
  The Hopkins Verbal Learning Test is a brief assessment of immediate recall, delayed recall and delayed recognition commonly used with populations with Alzheimer's disease, Huntington's disease and amnesic disorders. The maximum score for the test is 36 with scores below 14, indicating dementia. The minimum score is 0 and the maximum score is 36. A higher score indicates better working memory. The test takes about 5-10 minutes to take.
Change in Dual Tasking ability as measured by the Trail Making Test | Baseline, 24 weeks
  The Trail Making Test (TMT) is commonly used to screen for dementia by assessing the ability to think, reason, and remember. The score is how long it takes to complete the test. There is no minimal score, and the maximum score is 5 minutes. A lower the score the better the ability to reason and remember. The test takes about 7 minutes.
Change in cardiovascular fitness as measured by the Six-minute walk test. | Baseline, 24 weeks
  The six-minute walk test requires the subject to walk as far as possible in six minutes. The score is the distance traveled. The minimal score would be 0 and there is no maximum score. The further a person walks the better the cardiovascular condition. The test takes 6 minutes.
Change in neuromuscular performance as measured by 1-repetition maximum (1RM) | Baseline, 24 weeks
  Maximal load that can be lifted in one repetition (1RM) will be assessed for in both leg press and chest press exercises. The loads on the testing equipment will be increased over 5 to 7 testing sets. The persons 1RM will be the highest load the person can move through the range of motion of the exercise. There are no minimum or maximum scores for this test.
  The test typically takes 5 to 10 minutes. The higher the 1RM the stronger the person is.
Change in Concept Switching as measured by the Dimensional Card Sort test. | Baseline, 24 weeks
  The Dimensional Change Card Sort test is a measure of cognitive flexibility. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). "Switch" trials are also employed, in which the participant must change the dimension being matched. Scoring is based on a combination of accuracy and reaction time. Scores can range from 0-10. The higher the score, the better the capacity to switch from one concept to another. The test typically lasts four minutes.
Change in Congruent and Incongruent Responses as measured by the Flanker test | Baseline, 24 weeks
  The Flanker Test uses response inhibition to assess a subject's capacity to suppress incorrect responses within a particular context. The target (for this study an arrow) is flanked by non-target arrows that are either in the same direction as the target (congruent flankers), the opposite response (incongruent flankers), or to neither (neutral flankers). The minimum score is 0 and the maximum score is 10. A higher score indicates better accuracy. The test takes about 3 minutes.
Change in neuromuscular performance as measured by power production. | Baseline, 24 weeks
  This test measures the power a person can produce at maximal speed using a load of 50% of 1RM for the chest press and leg press. There are no minimum or maximum scores. The higher score is better. Power shows how fast a person can do work. The test typically takes about five minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neuromuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No